CLINICAL TRIAL: NCT06995547
Title: Digital Workflow Versus Functional Pick-up Techniques of Two- Implant Retained Mandibular Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Aya ebrahim elsayed elsayed elnagar, clinical demonstrator, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M36080622
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Occlusal Analysis
Keywords: CAD-CAM, implant, locator attachment, occlusense.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- functional pick up Group (Active Comparator)
  Interventions: Device: implant overdenture
- digital pick up Group (Active Comparator)
  Interventions: Device: implant overdenture

INTERVENTIONS:
Device: implant overdenture — Each patient will be receive two dental implants for overdenture fixation

SUMMARY:
The goal of this clinical trial] is to learn if digital pick up can affect occlusal forces on teeth in completely edentulous patients restored with digital complete overdenturs. The main question it aims to answer is:

Researchers will compare digital vs functional pick-up techniques to see if it affects occlusal force.

Participants will be asked to bite on digital articulating paper (occlusense).

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous, healthy firm mucosa without any remaining roots or jaw cysts. Maxillomandibular Angel's class I relationship with sufficient restorative space (minimum of 8.5 mm measured by using putty index). Sufficient residual alveolar bone quantity and quality class 1-3

Exclusion Criteria:

* Patients with systemic issues such as recent myocardial infarction, hepatic patients, bleeding disorders, autoimmune diseases like rheumatoid arthritis, hyperparathyroidism, uncontrolled diabetes mellitus, severe osteoporosis or cancer were excluded from the study. Also, patients with recent organ transplants, long-term corticosteroid use, radiotherapy, uncooperative patients with psychiatric disorders, heavy smokers, poor oral hygiene, and parafunctional habits were excluded

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
occlusal force analysis | twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah mohamed Ibrahim, assistant professor, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: No